CLINICAL TRIAL: NCT06880042
Title: COMPARISON OF EFFICACY AND SAFETY OF NARROWBAND UVB WITH 0.1% TACROLIMUS VS NARROWBAND UVB WITH 0.005% CALCIPOTRIOL IN TREATMENT OF VITILIGO
Acronym: NB-UVB
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dr ayesha wahid (Other Government)
Responsible Party: Sponsor-Investigator, Dr ayesha wahid, Awahid, Lahore General Hospital
Organization: Lahore General Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LGH
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-03

CONDITIONS: Vitiligo - Macular Depigmentation; Tacrolimus
Keywords: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Tacrolimus; calcipotriene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus (Active Comparator): Patient of Limited vitiligo less than 20% BSA will be treated with topical tacrolimus and narrowband UVB
  Interventions: Drug: Tacrolimus
- Calcipotriol (Active Comparator): Calcipotriol is a vitamin D analogue that will act as immunomodulator
  Interventions: Drug: Calcipotriol

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus is calcineurin inhibitor that will act as immunomodulator
  Arms: Tacrolimus
Drug: Calcipotriol — Calcipotriol is a vitamin D analogue that will act as immunomodulator
  Arms: Calcipotriol

SUMMARY:
Patient of stable and limited vitiligo less than 20% BSA will be recruited And evaluation of efficacy and safety of narrowband UVB with topical tacrolimus vs narrowband UVB and calcipotriol will be assessed

DETAILED DESCRIPTION:
Evaulation of efficacy and safety of narrowband uvb and tacrolimus and NBUVB and calcipotriol in patient if stable vitiligo with body surface area less than 20% It will be assessed by VASI score and VIisual analogie scale

ELIGIBILITY:
Inclusion Criteria:

- Localized vitiligo Age 15 to 70years Body surface upto 20% Stable more than 3 months

Exclusion Criteria:

* • Pregnant or lactating female patients.

  * Skin malignancy or any other malignant skin condition.
  * Photo induced or photo aggravated dermatosis like (SLE, photodermatitis, rosacea, psoriasis, pemphigus vulgaris) along with vitiligo.
  * Prior history of allergy to tacrolimus or calcipotriol.
  * Other form of treatment for vitiligo within at least 1 month.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
VASI improvement upto 50% | 3 months
  Improvement in VASI score upto 50%

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore general.hospital, Lahore, Punjab Province, Pakistan